CLINICAL TRIAL: NCT00438438
Title: "Interaction of Chronic Sleep Restriction and Circadian Misalignment on Sleep and Neuro-cognitive Performance"
Brief Title: Interaction of Chronic Sleep Restriction and Circadian Misalignment on Sleep and Neuro-cognitive Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth B. Klerman, Associate Professor, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 2200-100792
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Healthy
Keywords: forced desynchrony; circadian rhythms; sleep restriction; sleep homeostasis; neurobehavioral performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: forced desynchrony protocol with sleep restriction — Subjects are scheduled to live on a non-24 hour day. This separates the sleep-wake schedule from the near-24 hour circadian rhythm. This allows assessment of how circadian rhythms and the length-of-time awake contribute to sleepiness, alertness, and cognitive performance.

SUMMARY:
The primary objectives of the proposed experimental and modeling efforts are to quantify the influences of acute sleep deprivation (short-term homeostatic), chronic sleep restriction (long-term homeostatic), circadian rhythmicity, and their interactions on neurocognitive performance and to develop a new model of sleep homeostasis that can predict the effects of chronic sleep restriction. This model will be based on the underlying neuroanatomy and neurophysiology. This new model will facilitate optimization of human performance in operational settings, such as are seen in military operation and other work environments.

DETAILED DESCRIPTION:
This protocol involves a baseline period consisting of 14 hours of wakefulness and 10 hour nocturnal sleep episodes each 24 hours. This is followed by a forced desynchrony regimen spanning 21 calendar days and consisting of 12 cycles ("days") of a 42.85-hour wake:bedrest schedule. In each 42.85 hour cycle, there are 32.85 hours of scheduled wakefulness and 10 hour sleep opportunities. This will allow assessment of the independent contributions of circadian phase and homeostatic sleep pressure on sleep and neurobehavioral performance. This forced desynchrony regimen is followed by 10 recovery days consisting of 14 hours of wakefulness and 10 hour nocturnal sleep episodes each 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35 years old
* Medically healthy

Exclusion Criteria:

* Sleep disorder
* Psychiatric illness
* Chronic medical condition
* No prescription or Non-prescription medications

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Estimated)
Dates: Start 2006-04; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Sleep Stage | 38 days
Circadian Phase (melatonin rhythm) | 38 days
Psychomotor Vigilance Task | 38 days
Digit Symbol Substitution Task | 38 days
Addition Task | 38 days
Karolinska Sleepiness Scale | 38 days
Karolinska Drowsiness Test | 38 days
Mood Scales | 38 days
Flanker Task | 38 days
Multiple Object Tracking | 38 days

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth B Klerman, M.D., Ph.D., Principal Investigator — Brigham and Woman's Hospital; Charles A Czeisler, Ph.D., M.D., Principal Investigator — Brigham and Woman's Hospital
Locations (1):
- Brigham and Woman's Hospital, Boston, Massachusetts, United States